CLINICAL TRIAL: NCT01166347
Title: A Prospective, Randomized, Controlled, Un-blinded, Multi-Center Clinical Trial to Evaluate the HeartWare™ Ventricular Assist System (VAS) for Destination Therapy of Advanced Heart Failure
Brief Title: The HeartWare™ Ventricular Assist System as Destination Therapy of Advanced Heart Failure: the ENDURANCE Trial
Acronym: ENDURANCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HW004 ENDURANCE
Record Dates: First submitted 2010-07-16; First posted 2010-07-21 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HeartWare® VAS (Experimental): Implant of HeartWare® Ventricular Assist System
  Interventions: Device: HeartWare® VAS
- Control LVAD (Active Comparator): Implant of FDA-approved LVADs approved for destination therapy
  Interventions: Device: Control LVAD

INTERVENTIONS:
Device: HeartWare® VAS — The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
  Arms: HeartWare® VAS
Device: Control LVAD — Any FDA-approved LVAD for destination therapy.
  Arms: Control LVAD

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the HeartWare Ventricular Assist System in patients with chronic Stage D/ New York Heart Association (NYHA) Class IIIB/IV left ventricular failure who have received and failed optimal medical therapy, and who are ineligible for cardiac transplantation.

DETAILED DESCRIPTION:
The HeartWare Ventricular Assist System (VAS) is intended for use in patients with chronic Stage D/NYHA Class IIIB/IV left ventricular failure who have received and failed optimal medical therapy and who are ineligible for cardiac transplantation. The ENDURANCE clinical study is a prospective, randomized, unblinded, multi-center, non-inferiority evaluation of the HeartWare® VAS versus a control group consisting of any FDA-approved Left Ventricular Assist Device (LVAD) approved for destination therapy. Patients are randomized to HeartWare® VAS or control LVAD in a 2:1 ratio. Each patient receiving the HeartWare® VAS or control LVAD is followed to the primary endpoint at 2 years, with a subsequent follow-up period extending to 5 years post implant.

ELIGIBILITY:
Inclusion Criteria:

1. Must be ≥18 years of age at consent
2. Body Surface Area (BSA) ≥ 1.2 m2
3. Patients with advanced heart failure symptoms (New York Heart Association (NYHA) Class IIIB or IV) who are: (patient must meet one of the following) 3a. On optimal medical management, including dietary salt restriction and diuretics, for at least 45 out of the last 60 days and are failing to respond; or 3b. In NYHA Class III or NYHA Class IV heart failure for at least 14 days, and dependent on intra aortic balloon pump (IABP) for 7 days and/or inotropes for at least 14 days
4. Left ventricular ejection fraction ≤ 25%
5. LVAD implant is intended as destination therapy
6. Must be able to receive either the HeartWare® VAS or control LVAD
7. Female patients of childbearing potential must agree to use adequate contraceptive precautions for the duration of the study.
8. The patient or legally authorized representative has signed the informed consent form

Exclusion Criteria:

1. Body Mass Index (BMI) > 40
2. Existence of any ongoing mechanical circulatory support (MCS) other than an intra-aortic balloon pump (IABP)
3. Prior cardiac transplant.
4. History of confirmed, untreated abdominal or thoracic aortic aneurysm > 5 cm.
5. Cardiothoracic surgery within 30 days of randomization.
6. Acute myocardial infarction within 14 days of implant
7. Patients eligible for cardiac transplantation
8. On ventilator support for > 72 hours within the four days immediately prior to randomization and implant.
9. Pulmonary embolus within three weeks of randomization
10. Symptomatic cerebrovascular disease, stroke within 180 days of randomization or > 80% stenosis of carotid or cranial vessels.
11. Uncorrected moderate to severe aortic insufficiency. Correction may include repair or bioprosthesis at the time of implant.
12. Severe right ventricular failure as defined by the anticipated need for right ventricular assist device (RVAD) support or extracorporeal membrane oxygenation (ECMO) or right atrial pressure > 20 mmHg on multiple inotropes, right ventricular ejection fraction (RVEF) <15% or clinical signs
13. Active, uncontrolled infection diagnosed by a combination of clinical symptoms and laboratory testing.
14. Uncorrected thrombocytopenia or generalized coagulopathy (e.g., platelet count < 75,000, INR > 2.0 or PTT > 2.5 times control in the absence of anticoagulation therapy).
15. Intolerance to anticoagulant or antiplatelet therapies or any other peri- or postoperative therapy that the investigator may administer based upon the patient's health status.
16. Serum creatinine > 3.0 mg/dL within 72 hours of randomization or requiring dialysis (does not include use of ultra-filtration for fluid removal).
17. Specific liver enzymes [AST (SGOT) and ALT (SGPT)] > 3 times upper limit of normal within 72 hours of randomization.
18. A total bilirubin > 3 mg/dl within 72 hours of randomization, or biopsy proven liver cirrhosis or portal hypertension.
19. Pulmonary vascular resistance (PVR) is demonstrated to be unresponsive to pharmacological manipulation and the PVR > 6 Wood units.
20. Patients with a mechanical heart valve .
21. Etiology of heart failure is due to, or associated with, uncorrected thyroid disease, obstructive cardiomyopathy, pericardial disease, amyloidosis, active myocarditis or restrictive cardiomyopathy
22. History of severe Chronic Obstructive Pulmonary Disease (COPD) or severe restrictive lung disease
23. Participation in any other study involving investigational drugs or devices
24. Severe illness, other than heart disease, which would limit survival to < 3 years
25. Peripheral vascular disease with rest pain or ischemic ulcers of the extremities
26. Pregnancy
27. Patient unwilling or unable to comply with study requirements
28. Technical obstacles, which pose an inordinately high surgical risk, in the judgment of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2010-08; Primary Completion 2014-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis Pagani, MD, Principal Investigator — University of Michigan Hospital; Joseph Rogers, MD, Principal Investigator — Duke University
Locations (48):
- United States (48):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Hospital - Phoenix, Phoenix, Arizona
  - The University of Southern California, Los Angeles, California
  - Sharp Memorial, San Diego, California
  - Stanford University School of Medicine, Stanford, California
  - University of Colorado Hospital - Leprino, Aurora, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida - Gainesville, Gainesville, Florida
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - Tampa Transplant Institute/Tampa General Hospital, Tampa, Florida
  - The Emory Clinic Inc., Atlanta, Georgia
  - Saint Joseph Hospital of Atlanta, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - IU Health Methodist, Indianapolis, Indiana
  - Saint Vincent Health, Indianapolis, Indiana
  - Jewish Hospital, Louisville, Kentucky
  - John Ochsner Heart & Vascular Institute, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Abbott Northwestern, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. Mary's Hospital - Mayo, Rochester, Minnesota
  - Washington University/Barnes-Jewish Hospital, St Louis, Missouri
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - New York Presbyterian Hospital/Columbia, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas - South Western, Dallas, Texas
  - Texas Heart Institute, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - Innova Heart and Vascular Institute Research - Cardiac Vascular & Thoracic Surgery Associates, PC, Falls Church, Virginia
  - Sentara Norfolk, Norfolk, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Northwest Cardiothoracic &Transplant Surgeons, Spokane, Washington
  - Saint Luke's Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Result] Rogers JG, Pagani FD, Tatooles AJ, Bhat G, Slaughter MS, Birks EJ, Boyce SW, Najjar SS, Jeevanandam V, Anderson AS, Gregoric ID, Mallidi H, Leadley K, Aaronson KD, Frazier OH, Milano CA. Intrapericardial Left Ventricular Assist Device for Advanced Heart Failure. N Engl J Med. 2017 Feb 2;376(5):451-460. doi: 10.1056/NEJMoa1602954. PMID 28146651
- [Derived] Mahr C, McGee E Jr, Cheung A, Mokadam NA, Strueber M, Slaughter MS, Danter MR, Levy WC, Cheng RK, Beckman JA, May DM, Ismyrloglou E, Tsintzos SI, Silvestry SC. Cost-Effectiveness of Thoracotomy Approach for the Implantation of a Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):855-861. doi: 10.1097/MAT.0000000000001209. PMID 32740343
- [Derived] Silvestry SC, Mahr C, Slaughter MS, Levy WC, Cheng RK, May DM, Ismyrloglou E, Tsintzos SI, Tuttle E, Cook K, Birk E, Gomes A, Graham S, Cotts WG. Cost-Effectiveness of a Small Intrapericardial Centrifugal Left Ventricular Assist Device. ASAIO J. 2020 Aug;66(8):862-870. doi: 10.1097/MAT.0000000000001211. PMID 32740129
- See also: Intrapericardial Left Ventricular Assist Device for Advanced Heart Failure — http://www.nejm.org/doi/full/10.1056/NEJMoa1602954#t=articleTop

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five enrolled subjects were not randomized to a group due to lack of written insurance approval to receive the study device, death prior to randomization, prior screen failure (later improved), or withdrawal of consent.
Groups:
- HeartWare® Ventricular Assist System (VAS): HeartWare® Ventricular Assist System(VAS): The HeartWare® VAS is an implantable centrifugal pump that was designed to provide flows up to 10 L/min in a small device that is both lightweight and simple to use.
- Control Left Ventricular Assist Device (LVAD): Control Left Ventricular Assist Device (LVAD): Any Food and Drug Administration (FDA)-approved LVAD for destination therapy.
Period: Overall Study
Arm/Group | HeartWare® Ventricular Assist System (VAS) | Control Left Ventricular Assist Device (LVAD)
Started | 297 | 149
Completed | 295 | 148
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Only randomized subjects who successfully received an implant are included.
Groups:
- Total: Total of all reporting groups
Arm/Group | HeartWare® VAS | Control LVAD | Total
Number analyzed (Participants) | 297 | 148 | 445
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (11.60) | 66.2 (10.23) | 64.7 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 26 | 96
  Male | 227 | 122 | 349
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 15
  Not Hispanic or Latino | 288 | 142 | 430
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Black or African American | 66 | 32 | 98
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 228 | 115 | 343
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Stroke-Free Survival Probability for 2 Years Post Implant
Description: The primary endpoint of the trial is stroke-free survival at two years, defined as alive on the originally implanted device, electively transplanted or explanted due to patient recovery and free from disabling stroke (Modified Rankin Scale >=4). The Modified Rankin Scale is scored from 0 to 6, where 0 indicates an absence of symptoms and 6 indicates death. A score of 4 or higher indicates moderately severe or greater disability. Weibull model estimates of survival probability (shown as a percent of 100) are used.
Time Frame: Implant to 2 years
Population: Only randomized subjects who successfully received an implant are included.
Measure: Number; unit: Probabillity
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 297 | 148
Probabillity | 55.4 | 59.1
Statistical Analysis 1: Comparison: HeartWare® VAS vs Control LVAD; Primary endpoint is 2 year survival free from disabling stroke (Modified Rankin Scale >=4), death, exchange, explant due to device malfunction or urgent transplantation. Subjects who are electively transplanted or explanted due to recovery (no disabling stroke) must survive to 2 years post original implant to be considered a success; Test type: Non-Inferiority — The non-inferiority margin was 15%; p = 0.0110, Wald test; Difference in Percentages = 3.7, 95% CI 1-sided [upper limit 12.56] — Difference = Control - HeartWare

2. Secondary Outcome: Number of Participants With Bleeding
Description: Number of participants with bleeding, per Interagency Registry for Mechanically Assisted Circulatory Support (INTERMACS) definition. The event of bleeding is defined as: An episode of suspected internal or external bleeding that results in one or more of the following:
  1. Death,
  2. Re-operation,
  3. Hospitalization,
  4. Transfusion of red blood cells as follows:
  During first 7 days post implant
  * Adults (≥ 50 kg): ≥ 4U packed red blood cells (PRBC) within any 24 hour period during first 7 days post implant.
  After 7 days post implant
  * Any transfusion of packed red blood cells (PRBC) after 7 days following implant.
Time Frame: Implant to two years
Population: Only randomized subjects who successfully received an implant are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 297 | 148
Participants | 180 | 88
Statistical Analysis 1: Comparison: HeartWare® VAS vs Control LVAD; If non-inferiority is established for the primary endpoint, statistical testing for superiority and p-value estimation for the 3 secondary endpoints (incidence of bleeding, incidence of major infection, overall survival) will be performed in a pre-specified sequence and testing will continue at the nominal alpha level until the first non-significant result. This fixed sequence procedure strongly controls the family-wise error rate for the collection of the 3 secondary endpoints; Test type: Superiority; p = 0.5922, Regression, Logistic — If p<0.05, then the test is statistically significant; Treatment as the only independent variable; Difference in Percentages = 1.1, 95% CI 2-sided [-8.5 to 10.8] — Difference = HeartWare - Control

3. Secondary Outcome: Number of Participants With Major Infections
Description: Number of participants with major infections, per INTERMACS definition. A major infection is defined as: A clinical infection accompanied by pain, fever, drainage and/or leukocytosis that is treated by anti-microbial agents (non-prophylactic). A positive culture from the infected site or organ should be present unless strong clinical evidence indicates the need for treatment despite negative cultures. The general categories of infection include Localized non-device infection Percutaneous site and/or pocket infection Internal pump component, inflow or outflow tract infection Sepsis
Time Frame: Implant to two years
Population: Only randomized subjects who successfully received an implant are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 297 | 148
Participants | 206 | 92

4. Secondary Outcome: Overall Survival at 2 Years
Description: Overall survival is the probability (expressed as a percent of 100) did not died within 2 years post implant via the Kaplan-Meier method. Participants that did not died were censored at the time of last follow-up or 2 years post implant, whichever occurred first.
Time Frame: Implant to two years
Population: Only randomized subjects who successfully received an implant are included.
Measure: Number; unit: Probability
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 297 | 148
Probability | 60.7 | 67.6

5. Secondary Outcome: Number of Participants With Device Malfunctions
Description: Number of Participants with device malfunctions per INTERMACS definition. Device malfunction denotes a failure of one or more of the components of the Mechanical Circulatory Support Device (MCSD) system which either directly causes or could potentially induce a state of inadequate circulatory support (low cardiac output state) or death. The manufacturer must confirm device failure. A failure that was iatrogenic or recipient-induced will be classified as an Iatrogenic/Recipient-Induced Failure.
  Device failure should be classified according to which components fails as follows:
  1. Pump failure (blood contacting components of pump and any motor or other pump actuating mechanism that is housed with the blood contacting components).
  2. Non-pump failure (e.g., external pneumatic drive unit, electric power supply unit, batteries, controller, interconnect cable, compliance chamber)
Time Frame: Implant to two years
Population: Only randomized subjects who successfully received an implant are included.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 297 | 148
Participants | 93 | 38

6. Secondary Outcome: Health Status Change Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: Health Status change as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score. The KCCQ is a disease-specific patient-reported outcomes measure for patients with heart failure. It consists of 23 items, is comprised of 7 clinically relevant scales (Symptom Frequency, Symptom Burden, Symptom Stability, Physical Limitation, Social Limitation, Quality of Life, and Self-Efficacy), and yields 3 summary scores (Clinical Summary, Total Symptom, and Overall Summary Scores). Scale and summary scores range between 0 and 100, with higher scores indicating better health status (e.g., better functioning, fewer symptoms, better quality of life). The Overall Summary Score is calculated as the mean of the Physical Limitation, Total Symptom, Quality of Life and Social Limitation scores. A positive change in score from baseline indicates an improvement.
Time Frame: Change from baseline to 2 years
Population: Only randomized subjects who successfully received an implant are included. Subjects also had to reach the Month 24 visit and complete both the baseline and Month 24 assessments to be analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 138 | 76
Units on a scale | 30.2 (24.12) | 30.8 (28.81)

7. Secondary Outcome: Health Status Change Measured by EuroQol EQ-5D (Version 3L)
Description: The EuroQol-5D (version 3L) is a brief self-administered, validated instrument consisting of 2 parts. The second part consists of the EQ-5D general health status as measured by a visual analog scale (EQ-5D VAS). EQ-5D VAS measures the participant's self-rated health status on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state). An adjustment was done on the response where the scores were normalized based on this paper: Johnson JA, Coons SJ. Comparison of the EQ-5D and SF-12 in an adult US sample. Qual Life Res. 1998 Feb;7(2):155-66.
Time Frame: Change from baseline to 2 years
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 139 | 77
units on a scale | 1.7 (1.98) | 1.8 (2.23)

8. Secondary Outcome: Change in Functional Status Measured by New York Heart Association (NYHA) Class
Description: Change in Functional status, as measured by New York Heart Association (NYHA) class. There are 4 levels of NYHA:
  I (Mild): No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, or dyspnea.
  II (Mild): Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea.
  III (Moderate): Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV (Severe): Unable to carry out any physical activity without discomfort. Symptoms of cardiac insufficiency at rest. If any physical activity is undertaken, discomfort is increased. Improvement is defined as moving from a higher numerical NYHA level to a lower numerical NYHA level (e.g., IV to III).
Time Frame: Change from baseline to 2 years
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 152 | 84
Participants
  Worsened 1 NYHA Class | 2 | 0
  No Change in NYHA Class | 15 | 6
  Improved 1 NYHA Class | 39 | 19
  Improved 2 NYHA Classes | 63 | 40
  Improved 3 NYHA Classes | 33 | 19

9. Secondary Outcome: Change in Functional Status as Measured by 6-minute Walk
Description: Change in functional status, as measured by 6-minute walk test.
Time Frame: Change from baseline to 2 years
Population: Only randomized subjects who successfully received an implant are included. Subjects also had to reach the Month 24 visit and complete the assessment or indicate Not Completed to be analyzed at both the baseline and Month 24 visits. If the subject did not complete the assessment, a value of 0 was imputed.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 160 | 89
Meters | 95.6 (177.09) | 109.8 (181.34)

10. Secondary Outcome: Length of Initial Hospitalization
Description: Length of Initial Hospitalization post implant
Time Frame: Implant to the end of the initial hospitalization
Population: Only randomized subjects who successfully received an implant are included. Subjects are analyzed based on the device they actually received. Subjects who died while in the hospital or have a missing discharge date were not included.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 265 | 132
Days | 26.0 (20.52) | 25.0 (15.58)

11. Secondary Outcome: Number of Participants Who Had a Re-hospitalization
Description: Number of participants who had a re-hospitalization while on the device
Time Frame: Implant to two years
Population: Only randomized subjects who successfully received an implant are included. Subjects are analyzed based on the device they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 296 | 149
Participants | 249 | 118

12. Secondary Outcome: Duration of Re-hospitalization
Description: Duration of Re-hospitalization while on device
Time Frame: Implant to two years
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 241 | 118
Days | 44.1 (37.01) | 39.3 (33.77)

13. Secondary Outcome: Cause of Re-hospitalization
Description: Cause of Re-hospitalization while on device. The reason a participant may have been re-hospitalized was due to an adverse event, the need for an explant, or for various "Other" reasons.
Time Frame: Implant to two years
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | HeartWare® VAS | Control LVAD
Number analyzed (Participants) | 296 | 149
Participants
  Adverse Event | 241 | 107
  Explant | 33 | 28
  Other | 53 | 32

ADVERSE EVENTS:
Time Frame: The adverse events are summarized from the date of implant through 2 years while on the originally implanted device. Only randomized subjects who successfully received an implant are included. Subjects are analyzed based on the device they actually received.
Description: The Interagency Registry for Mechanically Assisted Circulatory Support (Intermacs) adverse event definitions are geared towards subjects who have a mechanical circulatory support device.
Arm/Group | HeartWare® VAS | Control LVAD
All-Cause Mortality (participants affected / at risk) | 116/296 | 48/149
Serious Adverse Events (participants affected / at risk) | 284/296 | 141/149
Other Adverse Events (participants affected / at risk) | 112/296 | 50/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=296) | Control LVAD (N=149)
Major Bleeding (Blood and lymphatic system disorders) | 170 (377) | 87 (189)
Cardiac Arrhythmia (Cardiac disorders) | 98 (153) | 55 (74)
Device Malfunction (Product Issues) | 71 (82) | 34 (37)
Hemolysis (Blood and lymphatic system disorders) | 25 (33) | 14 (15)
Hepatic Dysfunction (Hepatobiliary disorders) | 14 (14) | 11 (11)
Hypertension (Cardiac disorders) | 32 (39) | 18 (21)
Major Infection (Infections and infestations) | 185 (389) | 79 (145)
Myocardial Infarction (Cardiac disorders) | 4 (4) | 0 (0)
Neurological Dysfunction (Nervous system disorders) | 97 (140) | 25 (26)
Pericardial Fluid Collection (Cardiac disorders) | 8 (8) | 9 (9)
Psychiatric Episode (Psychiatric disorders) | 34 (36) | 10 (11)
Renal Dysfunction (Renal and urinary disorders) | 43 (52) | 17 (18)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 81 (109) | 36 (46)
Right Heart Failure (Cardiac disorders) | 99 (114) | 35 (40)
Arterial Non-CNS Thromboembolism (Vascular disorders) | 5 (6) | 3 (9)
Venous Thromboembolism (Vascular disorders) | 8 (11) | 5 (5)
Wound Dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Other Intermacs (General disorders) | 226 (724) | 107 (301)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HeartWare® VAS (N=296) | Control LVAD (N=149)
Major Bleeding (Blood and lymphatic system disorders) | 26 (33) | 9 (10)
Cardiac Arrhythmia (Cardiac disorders) | 22 (25) | 9 (9)
Device Malfunction/Failure (Product Issues) | 28 (42) | 5 (6)
Hypertension (Cardiac disorders) | 18 (23) | 8 (8)
Major Infection (Infections and infestations) | 54 (76) | 26 (40)
Psychiatric Episode (Psychiatric disorders) | 17 (19) | 7 (7)
Right Heart Failure (Cardiac disorders) | 19 (19) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In most cases, the contract allows the principal investigator to publish their data after the release of the multi-center publication (or one year after the conclusion of the study if no multi-center publication is submitted) following the sponsor review for (a) disclosure of confidential information, and (b) information that would impair the sponsor's ability to obtain patent protection.